CLINICAL TRIAL: NCT01307449
Title: Systems Biology of 23 Valent Pneumococcal Polysaccharide Vaccine (PNEUMOVAX®23) and 13-valent Pneumococcal Conjugate Vaccine (PREVNAR 13®)
Brief Title: Systems Biology of PNEUMOVAX®23 and PREVNAR 13®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Nadine Rouphael, MD, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00047973; U19AI090023 (NIH); IRB00078300 (Other: Emory University IRB)
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Pneumococcal Infection
Keywords: pneumococcal vaccine; immune responses
MeSH Terms: conditions — Pneumococcal Infections | interventions — Pneumococcal Vaccines; 23-valent pneumococcal capsular polysaccharide vaccine; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Older Group on PREVNAR (Experimental): Participants between the ages of 60-89 received PREVNAR
  Interventions: Biological: Prevnar
- Younger Group on PREVNAR (Experimental): Participants between the ages of 25-40 years received PREVNAR
  Interventions: Biological: Prevnar
- Older Group on PNEUMOVAX (Experimental): Participants between the ages of 60-89 received PNEUMOVAX
  Interventions: Biological: PNEUMOVAX
- Younger Group on PNEUMOVAX (Experimental): Participants between the ages of 25-40 years received PNEUMOVAX
  Interventions: Biological: PNEUMOVAX

INTERVENTIONS:
Biological: PNEUMOVAX — 1 dose of PNEUMOVAX
  Other Names: 23-valent polysaccharide pneumococcal vaccine
  Arms: Older Group on PNEUMOVAX; Younger Group on PNEUMOVAX
Biological: Prevnar — 1 dose of Prevnar
  Other Names: 13-valent pneumococcal conjugate vaccine
  Arms: Older Group on PREVNAR; Younger Group on PREVNAR

SUMMARY:
Vaccination is the most effective way of preventing infectious diseases. Despite the success of vaccines in general, vaccines induce diminished antibody responses and lower protection in the elderly in particular. This could be explained by a defect in the early responses of an ageing immune system. A better understanding of the basic immunological mechanisms that mediate vaccine efficacy is incomplete. Such information is critical and could greatly decrease both the cost and the time to new vaccine development particularly for the geriatric population.

In this trial, the investigators will study the immunologic differences of two FDA approved licensed pneumococcal vaccines between a younger and an older group. Twenty two healthy volunteers between the age of 25-40 and sixty six healthy volunteers between the ages of 60-89 will be enrolled in the study. Each participant in the study will be given one pneumococcal shot. Blood work will be obtained prior to vaccination, one day, three days, seven days, fourteen days, as well as one month and six months after vaccination. Throughout the duration of the study, the participants will be monitored for safety.

DETAILED DESCRIPTION:
RATIONALE: PCV13 [13-valent pneumococcal conjugate vaccine (Prevnar®13)] induces better functional immune responses when compared to PPV23 [23-valent pneumococcal polysaccharide vaccine (Pneumovax®23)] in older naïve adults. We hypothesize that this is due to intrinsic defects in innate responses that could explain the poor immunogenicity of PPV23 when compared to PCV13. Therefore, we propose to extensively study innate and adaptive immune responses generated after administration of either pneumococcal polysaccharide or conjugate vaccines in older adults.

STUDY DESIGN: Single center, open label study in which adult healthy volunteers will be vaccinated with either PPV23 or PCV13. Blood samples will be collected on Days D0 (at enrollment) and D1, D3, D7, D14, D30 and D180 post vaccination to study innate and adaptive immune responses.

Even though PPV23 and PCV13 are considered safe, volunteers will be asked to report any local or systemic AEs from Day 0 (vaccination) to Day 7 . Reactogenicity events will also be evaluated by injection site examination on visits at D0, D1, D3 and D7. Also volunteers are asked to report any local or systemic AEs for 30 days post vaccination and any SAEs for 180 days post vaccination. Volunteers are also asked to report local and systemic AEs developing the day of a blood draw.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and give informed consent.
2. Immunocompetent community dwelling subjects between the ages of ages of 25-40 and 60-89 years.

Exclusion Criteria:

1. Prior vaccination with pneumococcal vaccine.
2. Receipt of any of the following products:

   1. Blood products within 3 months prior to study entry or expected receipt at any time after study entry*.
   2. Any live virus vaccines within 4 weeks prior to study entry or expected receipt within 4 weeks after study entry*.
   3. Any inactivated vaccine within 2 weeks or expected receipt within 2 weeks after study entry*.
3. Presence of co-morbidities or immunosuppressive states such as:

   * Chronic medical problems including (but not limited to) insulin dependent diabetes, severe heart disease, severe lung disease, severe liver disease, cerebrospinal fluid leaks, severe kidney disease, autoimmune diseases, severe gastrointestinal diseases and grade 4 hypertension per CTCAE criteria** .
   * Alcohol, drug abuse or psychiatric conditions that in the opinion of the investigator would preclude compliance with the trial or interpretation of safety or endpoint data.
   * Impaired immune function or known chronic infections including, but not limited, to known HIV, hepatitis B or C; organ transplant; immunosuppression due to cancer; current and/or expected receipt of chemotherapy, radiation therapy, steroids*** (i.e., more than 20 mg of prednisone given daily or on alternative days for 2 weeks or more in the past 90 days , or high dose inhaled corticosteroids**** or any other immunosuppressive therapies (including anti-TNF therapy), functional or anatomic asplenia and congenital immunodeficiency.
4. Conditions that could affect the safety of the volunteers such as:

   o Severe reactions to prior vaccinations.

   o An allergy to any component of the study vaccines (phenol, aluminum, CRM197 protein, succinic acid, Polysorbate 80).
   * History of Guillain-Barré syndrome.
   * History of bleeding disorders.
5. Volunteers with any acute illness* including, but not limited to, - fever (> 100.4 F [> 38 C], regardless of the route) within 3 days prior to study entry.
6. Volunteers with social conditions or occupational conditions or any condition that in the opinion of the investigator might interfere with compliance with the study and vaccine evaluation.
7. Pregnant or breast feeding or women expected to conceive within 30 days after vaccination *****

   * An individual who initially is excluded from study participation based on one or more of the time-limited exclusion criteria (e.g., acute illness, receipt or expected receipt of live or inactivated vaccines ) may be reconsidered for enrollment once the condition has resolved as long as the subject continues to meet all other entry criteria.

     * Grade 4 hypertension per CTCAE criteria is defined as Life threatening consequences(e.g., malignant hypertension, transient or permanent neurologic deficit, hypertensive crisis) urgent intervention indicated. ***Subjects receiving > 20 mg/day of prednisone or its equivalent daily or on alternate days for more than 2 weeks may enter the study after therapy has been discontinued for more than 3 months.

       * High dose ICS is defined as: > 960 mcg/day of beclomethasone dipropionate or equivalent ***** Women of child-bearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for ≥1 year) must agree to practice adequate contraception that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, and licensed hormonal methods for 30 days before and 30 days after receiving PPV23 or PCV13.

Ages: 25 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Hope Clinic of the Emory Vaccine Center, Decatur, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Older Group (60-89) PNEUMOVAX: Older Group (60-89) receiving single dose of PNEUMOVAX
- Older Group (60-89) PREVNAR: Older Group (60-89) receiving single dose of PREVNAR
- Younger Group (25-40) PNEUMOVAX: Younger Group (25-40) receiving single dose of PNEUMOVAX
- Younger Group (25-40) PREVNAR: Younger Group (25-40) receiving single dose of PREVNAR
Period: Overall Study
Arm/Group | Older Group (60-89) PNEUMOVAX | Older Group (60-89) PREVNAR | Younger Group (25-40) PNEUMOVAX | Younger Group (25-40) PREVNAR
Started | 33 | 33 | 11 | 11
Completed | 32 | 33 | 11 | 11
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Older Group (60-89) PNEUMOVAX | Older Group (60-89) PREVNAR | Younger Group (25-40) PNEUMOVAX | Younger Group (25-40) PREVNAR | Total
Number analyzed (Participants) | 33 | 33 | 11 | 11 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 11 | 11 | 36
  >=65 years | 27 | 25 | 0 | 0 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 7 | 4 | 47
  Male | 15 | 15 | 4 | 7 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 4 | 5 | 22
  White | 24 | 23 | 6 | 6 | 59
  More than one race | 1 | 3 | 0 | 0 | 4
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 11 | 11 | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Innate Immunity Signatures That Correlate With the Quality of Antibodies After PNEUMOVAX and PREVNAR - Monocyte Module M4.15
Description: Expression of select gene modules reporting on innate and adaptive responses in young and elderly vaccine recipients. Gene expression was compared between pre-vaccination baseline and post-vaccination day 7 for each subject. The number of subjects with significant (by FDR < 0.05) positive enrichment of Monocyte Module M4.15 is reported.
Time Frame: Day 7
Population: One of the subjects in Young Pneumovax group is missing the baseline (day 0) sample, which makes the analysis impossible. RNA was never isolated from this time point. The participant has completed the rest of the visits, but these samples can't be used for the analysis in the absence of baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Older Group (60-89) on PNEUMOVAX: Participants between the ages of 60-89 received single dose of PNEUMOVAX
- Older Group (60-89) on PREVNAR: Participants between the ages of 60-89 received single dose of PREVNAR
- Younger Group (25-40) on PNEUMOVAX: Participants between the ages of 25-40 years received single dose of PNEUMOVAX
- Younger Group (25-40) on PREVNAR: Participants between the ages of 25-40 years received single dose of PREVNAR
Arm/Group | Older Group (60-89) on PNEUMOVAX | Older Group (60-89) on PREVNAR | Younger Group (25-40) on PNEUMOVAX | Younger Group (25-40) on PREVNAR
Number analyzed (Participants) | 33 | 33 | 10 | 11
Participants | 1 | 2 | 0 | 2

2. Primary Outcome: Number of Participants With Innate Immunity Signatures That Correlate With the Quality of Antibodies After PNEUMOVAX and PREVNAR - Monocyte Module M11
Description: Expression of select gene modules reporting on innate and adaptive responses in young and elderly vaccine recipients. Gene expression was compared between pre-vaccination baseline and post-vaccination day 7 for each subject. The number of subjects with significant (by FDR < 0.05) positive enrichment of Monocyte Module M11 is reported.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Older Group (60-89) on PNEUMOVAX | Older Group (60-89) on PREVNAR | Younger Group (25-40) on PNEUMOVAX | Younger Group (25-40) on PREVNAR
Number analyzed (Participants) | 33 | 33 | 10 | 11
Participants | 1 | 5 | 0 | 3

3. Primary Outcome: Number of Participants With Innate Immunity Signatures That Correlate With the Quality of Antibodies After PNEUMOVAX and PREVNAR - Monocyte Module M73
Description: Expression of select gene modules reporting on innate and adaptive responses in young and elderly vaccine recipients. Gene expression was compared between pre-vaccination baseline and post-vaccination day 7 for each subject. The number of subjects with significant (by FDR < 0.05) positive enrichment of Monocyte Module M73 is reported.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Older Group (60-89) on PNEUMOVAX | Older Group (60-89) on PREVNAR | Younger Group (25-40) on PNEUMOVAX | Younger Group (25-40) on PREVNAR
Number analyzed (Participants) | 33 | 33 | 10 | 11
Participants | 0 | 3 | 0 | 2

4. Secondary Outcome: Number of Participants With Specific B Cell Responses at Day 7 That Correlate With the Innate Immune Signatures After PNEUMOVAX and PREVNAR - B Cell Module S3
Description: Expression of select B cell modules was compared between pre-vaccination baseline and 7 days post-vaccination for each subject individually. The number of subjects with significant (by FDR < 0.05) positive enrichment of B cell module S3 is reported.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Older Group (60-89) on PNEUMOVAX | Older Group (60-89) on PREVNAR | Younger Group (25-40) on PNEUMOVAX | Younger Group (25-40) on PREVNAR
Number analyzed (Participants) | 33 | 33 | 10 | 11
Participants | 9 | 10 | 7 | 8

5. Secondary Outcome: Number of Participants With Specific B Cell Responses at Day 7 That Correlate With the Innate Immune Signatures After PNEUMOVAX and PREVNAR - B Cell Module M156.0
Description: Expression of select B cell modules was compared between pre-vaccination baseline and 7 days post-vaccination for each subject individually. The number of subjects with significant (by FDR < 0.05) positive enrichment of B cell module M156.0 is reported.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Older Group (60-89) on PNEUMOVAX | Older Group (60-89) on PREVNAR | Younger Group (25-40) on PNEUMOVAX | Younger Group (25-40) on PREVNAR
Number analyzed (Participants) | 33 | 33 | 10 | 11
Participants | 28 | 25 | 9 | 9

6. Secondary Outcome: Number of Participants With Specific B Cell Responses at Day 7 That Correlate With the Innate Immune Signatures After PNEUMOVAX and PREVNAR - B Cell Module M156.1
Description: Expression of select B cell modules was compared between pre-vaccination baseline and 7 days post-vaccination for each subject individually. The number of subjects with significant (by FDR < 0.05) positive enrichment of B cell module M156.1 is reported.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Older Group (60-89) on PNEUMOVAX | Older Group (60-89) on PREVNAR | Younger Group (25-40) on PNEUMOVAX | Younger Group (25-40) on PREVNAR
Number analyzed (Participants) | 33 | 33 | 10 | 11
Participants | 32 | 30 | 10 | 11

ADVERSE EVENTS:
Time Frame: 6 months follow up (started at baseline)
Groups:
- Older Group (60-89) PNEUMOVAX: Participants between the ages of 60-89 received single dose of PNEUMOVAX
- Older Group (60-89) PREVNAR: Participants between the ages of 60-89 received single dose of PREVNAR
- Younger Group (25-40) PNEUMOVAX: Participants between the ages of 25-40 years received single dose of PNEUMOVAX
- Younger Group (25-40) PREVNAR: Participants between the ages of 25-40 years received single dose of PREVNAR
Arm/Group | Older Group (60-89) PNEUMOVAX | Older Group (60-89) PREVNAR | Younger Group (25-40) PNEUMOVAX | Younger Group (25-40) PREVNAR
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 3/33 | 2/33 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/33 | 0/33 | 0/11 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Older Group (60-89) PNEUMOVAX (N=33) | Older Group (60-89) PREVNAR (N=33) | Younger Group (25-40) PNEUMOVAX (N=11) | Younger Group (25-40) PREVNAR (N=11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lynch syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer recurrence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Older Group (60-89) PNEUMOVAX (N=33) | Older Group (60-89) PREVNAR (N=33) | Younger Group (25-40) PNEUMOVAX (N=11) | Younger Group (25-40) PREVNAR (N=11)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT01307449/Prot_SAP_000.pdf